CLINICAL TRIAL: NCT06717152
Title: A Randomized, Double-masked, Parallel, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of SJP-0132 Eye Drops Compared With Placebo in Chinese Patients With Dry Eye Disease
Brief Title: Efficacy and Safety of SJP-0132 Eye Drops in Chinese Patients With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Senju Pharmaceutical Science & Technology (Beijing) Co., Ltd. (Industry)
Collaborators: Senju Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJP-0132/3-03; CTR20244132 (Registry Identifier: Chinadrugtrials)
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SJP-0132 (Experimental): The participants receive placebo for 2 weeks in run-in period, then SJP-0132 for 8 weeks in treatment period.
  Interventions: Drug: SJP-0132; Drug: Placebo
- Placebo (Placebo Comparator): The participants receive placebo for 2 weeks in run-in period, then placebo for 8 weeks in treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SJP-0132 — Aqueous eye drop, one drop each time and four times each day, 8 weeks in treatment period in SJP-0132 group.
  Arms: SJP-0132
Drug: Placebo — Aqueous eye drop, one drop each time and four times each day, 2 weeks in run-in period in both groups and 8 weeks in treatment period in placebo group.

SUMMARY:
This study will evaluate the safety and efficacy of SJP-0132 in Chinese Patients with Dry Eye.

Patients will be randomly assigned to receive either SJP-0132 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 70 at the time of the informed consent
* Outpatient patients
* The patient's self-described dry eye symptom is more than 6 months or has the clinical diagnosis certificate of dry eye in the past 6 months at the time of the informed consent
* Tear film break-up time of <= 5 seconds at the beginning of screening and treatment period

Exclusion Criteria:

* Patients who have previously used SJP-0132 eye drops
* Patients who participated in or are currently participating in or planned to participate in other clinical studies within three months prior to the start of the screening period
* Patients who plan to wear corneal contact lenses between the beginning of the screening period and the end of the treatment period
* Patients who have undergone eye surgery (including laser surgery) or planned to undergo any eye surgery during the study period within one year prior to the beginning of the corneal transplantation surgery or screening period
* Any ophthalmic disease except for the dry eye (including eyeball or periocular infection, allergic or proliferative eye disease) is present at the beginning of the screening period and at the beginning of the treatment period. However, it does not include chronic eye disease patients who do not need treatment and may not become worse before the end of the treatment period
* Have known history of hypersensitivity or serious adverse reaction to any of the study drug ingredients
* Patients suffering from serious cardiovascular, respiratory, endocrine, digestive, urinary, blood, neurological, mental, ocular or peripheral malignancies (cured in or at the beginning of the screening period but not exceeding five years), at the beginning of screening and treatment period
* A patient at the beginning of screening and at treatment period who has a positive blood serum pregnancy test result or is in lactation, or a female patient who has planned pregnancy during the study period or has fertility but is unable to use effective contraception during the study period, or a female partner of a male patient who is unable to use effective contraception during the study
* Patients identified at the beginning of screening and treatment period as researchers, research coordinators, researchers and immediate relatives of the persons referred to above
* At the beginning of the screening and treatment period, investigators determine that patients who were unable to comply with the requirements of the program or were unable to come to hospital on schedule (e.g. patients who planned to travel or stay in the field during the period prior to the end of the treatment period)
* At the beginning of the screening and treatment period, investigators decide that the patients who were not suitable for the trial were not suitable for the other reasons
* Meet the other protocol-specified exclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Corneal Fluorescein Staining (CFS) Score at Total Zone | Day 29
  CFS score ranged from 0 to 5, where '0' represents no fluorescein staining, and '5' represents severe staining on the cornea. The higher scores mean worse outcomes.
Change From Baseline in Eye Dryness Symptom (VAS) | Day 8
  Visual analog scale (VAS): "0" mean none, and "100" mean the worst imaginable for the symptom question.

SECONDARY OUTCOMES:
Change From Baseline in Corneal Fluorescein Staining (CFS) Score at Total Zone | Day 8, 15, 57
  CFS score ranged from 0 to 5, where '0' represents no fluorescein staining, and '5' represents severe staining on the cornea. The higher scores mean worse outcomes.
Change From Baseline in Corneal Fluorescein Staining (CFS) Score in Each Zone (central, superior, temporal, nasal, and inferior) | Day 8, 15, 29, 57
  CFS score ranged from 0 to 5, where '0' represents no fluorescein staining, and '5' represents severe staining on the cornea. The higher scores mean worse outcomes.
Change From Baseline in Conjunctival Fluorescein Staining Score in Each Zone (temporal, temporal superior, temporal inferior, nasal superior, nasal inferior, and nasal) | Day 8, 15, 29, 57
  Conjunctival Fluorescein Staining score ranged from 0 to 5, where '0' represents no fluorescein staining, and '5' represents severe staining on the conjunctiva. The higher scores mean worse outcomes.
Change From Baseline in Symptoms Score (VAS) | Day 8, 15, 29, 57
  Visual analog scale (VAS): "0" mean none, and "100" mean the worst imaginable for the symptom question. VAS of Eye Dryness Symptom on Day 8 is excluded.
Change From Baseline in DEQ-5 Score | Day 29, 57
  The participants rated the frequency on a scale of 0 (never) to 4 (constant) with which they have experienced 3 symptoms (watery eyes, discomfort and dryness). The participant was also asked to rate the intensity of discomfort and dryness on a scale of 0 (never have it) to 5 (very intense). Total DEQ-5 score was the sum of scores for frequency and intensity of dryness and discomfort plus frequency of watery eyes. Maximum score is 22. Higher scores mean a worse outcome.
Change From Baseline in DEQS Score | Day 8, 15, 29, 57
  The DEQS score is composed of three categories of questions: questions about eye symptoms (6 questions), questions about the impact on daily life (9 questions), and question on general status (1 question). The questions regarding eye symptoms and the impact on daily life are scored in terms of their frequency and degree. The frequency is rated on a scale of 0 (never) to 4 (always) and the degree on a scale of 1 [hardly bothered me (not very bothersome)] to 4 [bothered me very much (very bothersome)]. The overall assessment is given on a scale of 1 (extremely good) to 6 (extremely bad). Maximum score is 100. The higher the score, the more severe the subjective symptoms of dry eye.
Change From Baseline in Symptom Diary Score | Day 8, 15, 29, 57
  The participants self-assess their dry eye symptoms using a diary. The scores are divided into several levels, ranging from 'not bothersome' to 'very troublesome,' with higher levels indicating worse symptoms.
Change From Baseline in Tear Film Break-up Time | Day 8, 15, 29, 57
  Tear film break-up time is the time taken for the first dry spot to appear on the cornea after a complete blink.
Change From Baseline in Tear Secretion | Day 29, 57
  The Schirmer's Test I method is used to measure tear secretion. The amount of tear secretion for 5 minutes is measured with a graduated Schirmer's test strip without topical ocular anesthetics. The longer the wetted portion of the test strip, the higher the tear secretion.

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Omatsu, Study Director — Senju Pharmaceutical Co., Ltd.
Locations (35):
- China (35):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xiamen Eye Center of Xiamen University, Xiamen, Fujian
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong, Shantou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Henan Eye Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - The Fourth Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Eye Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Norman Bethune Hospital of Jilin University, Changchun, Jilin
  - Dalian No.3 People's Hospital, Dalian, Liaoning
  - The Fourth People's Hospital of Shenyang, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Eye Hospital, Jinan, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - The first people's hospital of Xian Yang, Xianyang, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Ophthalmology Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo Eye Hospital, Ningbo, Zhejiang
  - Eye Hospital, WMU, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No